CLINICAL TRIAL: NCT05749679
Title: Prevention of NEphronic PErt in People With Type 2 DIABETIC Disease Followed in General Practice
Brief Title: Prevention of Renal Failure in People Followed for Type 2 Diabetes in General Practice
Acronym: PENEDIAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021_0864; 2022-A01698-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Renal Insufficiency and Diabetes Mellitus
Keywords: diabetes mellitus, type 2; kidney diseases; primary care; prevention; early diagnosis
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus; Diabetes Mellitus, Type 2; Kidney Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Physicians participating will receive training on renal failure in type 2 diabetes and on measures to reduce nephron loss
  Interventions: Other: training and audit
- Routine care (Sham Comparator)
  Interventions: Other: Routine care

INTERVENTIONS:
Other: training and audit — An evaluation of the practices with clinical audit before and after the management will be carried out.Every 3 months for 2 years, the investigating physicians of the intervention group will report for these patients the modifications or cessation of treatment, modification or implementation of interventions such as physical activity or implementation of nutritional modifications. Physician investigators will be asked to report any occurrence of adverse events to their regional pharmacovigilance centers.10 possible actions to be deployed :
  1. Hygienic and dietary measures
  2. Physical activity
  3. Smoking cessation
  4. Avoidance of nephrotoxic substances
  5. Treatment of hypertension
  6. Proteinuria reduction
  7. Oral antidiabetics; choice
  8. Optimal HBA1c
  9. Statin
  10. Compliance
  Arms: Training
Other: Routine care — Physicians in the "control" group will receive training on the study procedures. An evaluation of practices with a clinical audit before and after the treatments will be carried out. Every 3 months for 2 years, the investigating physicians in the control group will report for these patients the modifications or cessation of treatment, the modification or implementation of interventions such as physical activity or the implementation of modifications in terms of nutrition. The investigating physicians will be asked to report any occurrence of adverse events to their regional pharmacovigilance centers. Physician investigators in the control group will continue their care as usual.
  Arms: Routine care

SUMMARY:
This work will make it possible to identify the nephron loss of type 2 diabetic patients in the western region and to better define in general practice the impact of the elements put in place to reduce this loss and to raise awareness of the importance of these measures through training in comparison with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting his or her investigating general practitioner
* 50 years old or more
* type 2 diabetic for more than 5 years, with a GFR lower than 90 ml/mn and higher than 45 ml/mn (stage 2 and 3a of renal failure) and a nephron loss calculated on the average of the two previous years, higher than 3 ml/mn/year
* a microalbuminuria > 30 mg/gr of creatinuria.
* Having declared the investigator as the treating physician

Exclusion Criteria:

* Patient under 50 years of age Patients who do not agree to the use of their data (refusal of consent) or are unable to give consent (dementia, other) Patients with other types of diabetes Patients with renal failure other than diabetic or hypertensive glomerulopathy Patients unable to give consent Patients who do not understand the French language Patients with less than 3 months of planned follow-up Patients with a barrier to follow-up Patients undergoing dialysis, transplantation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in annual glomerular filtration rate (GFR) slope | Every 3 months during 2 years
  the annual glomerular filtration rate (GFR) slope calculated as the difference between the estimated loss over the two years before inclusion (N-2) and the estimated annual loss over the follow-up years after inclusion.

SECONDARY OUTCOMES:
Audit of clinical practices | before randomization, at 6 months and 24 months in the 2 groups
Cumulative incidence of unscheduled hospitalizations for all reasons at 2 years from the start of care in the intervention group compared to the control group | At 2 years (the end of the study)
change of Albuminuria | at baseline and every 3 months during the 2-year follow-up.